CLINICAL TRIAL: NCT06867328
Title: Comparison of Platelet-Rich Plasma Dressing and Normal Saline Dressing for Wound Healing in Patients With Chronic Diabetic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulab Devi Hospital (Other)
Responsible Party: Principal Investigator, Adeel Ahmed, Principal Investigator, Gulab Devi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GulabDeviH
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Wounds; Diabetic Ulcers
Keywords: Platelet-Rich Plasma (PRP); Normal Saline Dressing; Diabetic Ulcers; Chronic Wounds
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group PRP Dressing (Experimental): Patients in this group will receive platelet-rich plasma (PRP) dressing, which involves the application of autologous PRP to the chronic diabetic wound site. PRP will be prepared from the patient's own blood and applied twice weekly after wound debridement.
  Interventions: Procedure: Platelet-Rich Plasma (PRP) Dressing
- Group Normal Saline Dressing (Active Comparator): Patients in this group will receive normal saline dressing, which consists of cleansing the wound with normal saline followed by application of sterile gauze. This will be performed twice weekly after wound debridement.
  Interventions: Procedure: Normal Saline Dressing

INTERVENTIONS:
Procedure: Platelet-Rich Plasma (PRP) Dressing — * PRP will be prepared by centrifugation of 20 mL venous blood with an anticoagulant.
  * The extracted PRP will be applied twice weekly to the wound.
  * A sterile gauze will be placed over the wound after PRP application.
  * Treatment will continue for up to 6 weeks or until wound healing is achieved.
  Arms: Group PRP Dressing
Procedure: Normal Saline Dressing — Wound will be cleansed with normal saline and covered with sterile gauze.
  * Dressing changes will be done twice weekly following wound debridement.
  * Treatment will continue for up to 6 weeks or until wound healing is achieved.
  Arms: Group Normal Saline Dressing

SUMMARY:
Chronic diabetic wounds are a major health concern, often taking a long time to heal and increasing the risk of complications like infections and amputations. This study aims to compare the effectiveness of Platelet-Rich Plasma (PRP) Dressing versus Normal Saline Dressing in the treatment of chronic diabetic wounds. PRP is a treatment derived from the patient's own blood that contains growth factors, which may accelerate wound healing.

Participants with chronic diabetic wounds will be randomly assigned to receive either PRP dressing or normal saline dressing. The study will measure the rate of wound healing and the time taken to achieve complete healing in both groups. It is hypothesized that PRP dressing will lead to faster and more effective wound healing compared to normal saline dressing.

Findings from this research could help improve wound care strategies for diabetic patients and provide evidence for a more effective treatment approach in clinical practice.

DETAILED DESCRIPTION:
After obtaining approval from the institutional review board and obtaining informed consent from study participants, all patients fulfilling the inclusion criteria were included in the study from the surgery indoor department of Gulab Devi Hospital, Lahore. Baseline characteristics, including age (in years), gender (male/female), and history of comorbidities (hypertension/ischemic heart disease/smoking), were assessed by reviewing previous medical records and taking a detailed history. The duration of diabetes (in years), duration of the wound (weeks), size of the wound (measured using a millimeter scale along the longest axis), and class of chronic diabetic wound (III/IV) were documented.

After wound debridement, patients were randomized into two equal groups by block randomization as follows:

Group A: Patients were managed with normal saline dressing. Group B: Patients were managed with PRP dressing. In this technique, the wound was washed with normal saline, and platelet-rich plasma (prepared from the patient's own blood by the hematology department) was injected into the surrounding wound area twice weekly, followed by the placement of a gauze over it.

Dressing was continued for a period of 6 weeks or until wound healing was achieved, whichever was shorter. To assess healing, all patients in both groups were followed up weekly until 6 weeks (study endpoint). The duration required to achieve wound healing was also documented. Additionally, 6 weeks post-therapy, wound size was reassessed. In cases of non-healing, alternative therapy was provided based on the wound condition and the consultant surgeon's advice. All data were recorded in a predesigned proforma and kept confidential.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* Either male or female.
* Chronic diabetic wound.
* Wagner class III and IV.

Exclusion Criteria:

* Wound sustained < 6 weeks from time of presentation.
* Previous history of PRP dressing use, assessed by reviewing previous medical records.
* History of hypersensitivity to PRP, assessed by reviewing previous medical records.
* Burn injury, assessed by reviewing previous medical records.
* Class I, II and V.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Wound Healing | Evaluated weekly for up to 6 weeks
  Wound healing will be assessed based on the formation of pinkish granulation tissue completely covering the wound. The healing status will be determined by a consultant surgeon through visual inspection.

SECONDARY OUTCOMES:
Duration to Achieve Wound Healing | Measured at the end of 6 weeks or at the point of complete wound healing, whichever occurs first.
  The duration required for complete wound healing (formation of granulation tissue covering the entire wound) will be recorded in weeks for each patient in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulab Devi Chest Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No